CLINICAL TRIAL: NCT06524700
Title: Pectopexy Autologous Vs Mesh
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Armed forces hospital wadi aldwaser (Unknown)
Responsible Party: Principal Investigator, Hamdy Ahmed Saaid, Fellow, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAGVM
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Uterine Prolapse; Vault Prolapse, Vaginal
Keywords: vault; uterine; prolapse
MeSH Terms: conditions — Uterine Prolapse; Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator)
  Interventions: Procedure: pectopexy mesh
- B (Active Comparator)
  Interventions: Procedure: pectopexy autologous

INTERVENTIONS:
Procedure: pectopexy mesh — pectopexy with mesh
  Arms: A
Procedure: pectopexy autologous — pectopexy using autologous graft
  Arms: B

SUMMARY:
prospective comparative study describing using autologous graft for uterine- vault - cervical suspension vs mesh in treatment of apical prolapse

ELIGIBILITY:
Inclusion Criteria:

uterine - vault prolapse

-

Exclusion Criteria:

* previous vaginal repair for uterine or vaginal prolapse previous suspension procedures for apical prolapse

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
POP-Q | 3 month
  assesment of degree of prolapse correction after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Saaid, Study Chair — UROGYNECOLOGY UNIT
Locations (2):
- Urogynecology Unit, Cairo, Cairo Governorate, Egypt
- Armed forces Hospital Wadi Aldwaser, Riyadh, Wadi Aldwaser, Saudi Arabia